CLINICAL TRIAL: NCT06740318
Title: Recompensation in Alcohol Related Hepatitis- A Prospective Cohort With Alcohol Cessation
Brief Title: Recompensation in Alcohol Related Hepatitis
Acronym: A-HEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nina Kimer (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Sponsor-Investigator, Nina Kimer, MD, PhD, Associate Professor, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24040990
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Alcoholic Hepatitis (AH)
Keywords: alcohol use disorder; motivational enhancement therapy; metabolomics; incidence cohort; alcohol related hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic; Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Motivational enhancement therapy in three sessions within three months from diagnosis are applied in addition to standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Standard of Care: medical treatment of alcohol use disorder and motivational enhacement therapy, three interviews within three months.
  Interventions: Other: Motivational enhancement therapy

INTERVENTIONS:
Other: Motivational enhancement therapy — The intervention consists of three motivational interviews with the focus to enhance the participants motivation to enter treatment of alcohol use disorder. the interviews are structured and based on the model Motivational enhancement therapy.

SUMMARY:
Genetic activity and metabolic changes may be part of the pathogenesis in alcohol related hepatitis. We do not know exactly how alcohol cessation affects liver functions and metabolism.

The aim of this study is to assess the impact of alcohol cessation in patients with alcohol related hepatitis and gain knowledge of the metabolic and genetic functions of the liver during remission and recompensation from alcohol related hepatitis.

The study will assess

1. The effect of alcohol cessation on the liver.
2. The biological mechanisms involved in healing after alvohol-cessation
3. The effect of motivational enhcament therapy in alcohol cessation after alcohol related hepatitis.
4. The metabolic changes of lipids and proteins in the liver Participants are offered motivational enhancement therapy and standard of care.

DETAILED DESCRIPTION:
In a prospective incidence cohort study participants will be followed from diagnosis of Alcohol related Hepatitis (AH) until death or withdrawal from the cohort.

Participants will be included consecutively within one month of diagnosis.

All persons diagnosed with AH, and all patients with a debut of AH during admission, regardless of the reason for admission, are eligible for inclusion.

The study does not compromise diagnostics or treatment of AH, cirrhosis or comorbidities.

Inclusion criteria are: clinical suspicion of AH, supported by biochemistry (bilirubin 50 mmol/l or higher) and ultrasound or other imaging techniques; informed written consent.

Exclusion criteria are: People where the diagnosis of AH is questioned with reasonable doubt; withdrawal of informed consent; persons eligible for inclusion where the investigational program is delayed or not initiated within two months after the diagnosis of suspected AH; Persons with hepatocellular carcinoma.

Participants referred to the Gastro Unit for either admission or the out-patient clinic will be offered inclusion.

Alcohol cessation intervention:

All patients with AH treated in the Gastro Unit, AHH and hence, all participants in the study will be offered standard of care, including nutritional supplements, supportive care and medical treatment of complications or comorbidities. Support to alcohol cessation including medical treatment of withdrawal symptoms and craving, and one to three structured motivational interviews will be offered in the first 3 months after admission, as well as referral to municipal offers of alcohol treatment.

Data from patient journals:

Information from the patient records will be retrieved as:

Dates and length of hospitalizations; Reason for hospitalizations; Diagnoses; Biochemistry; Results from endoscopic procedures.

Data and personal information are registered and monitored after current Danish legislation, The Data Protection Act, and as stated by the Data Protection Regulation.

Quality of life and Health Questionnares regarding Quality of life and self-percieved health including mental health is applied in the study. The aim is to investigate the potential benefits of alcohol-cessation on quality of life and self-perceived health, including mental health. If a participant indicates signs of severe depression, referral to relevant institutions will be initiated, following national guidelines for depression.

Genetic analyses Genotyping will be performed with a GWAS-chip (i.e. targeted genomic mapping) using Illumina Exomechip enriched for protein-changing, large-effect variants. Ultra-rare variants (<1/1000) will not be captured. The results will be used to test the potential clinical value of genetic risk profiling in combination with clinical data. Genomic analysis comprises common variants and polygenic risk score profiling on common variants.

Proteomics, lipidomics and transcriptomics:

Preparation of samples and liquid chromatography and mass spectrometry (LC/MS) analysis will follow technologies previously described. The field of proteomics is rapidly evolving, and methods may be subject to adaptations to secure quality, relevance and the best prizes for the analysis.

We will analyze plasma proteomics datasets with Spectronaut v.15.4 . A previously generated deep fractionated plasma data-dependent acquisition (DDA) library is used in the targeted analysis of data independent application data against the human reference proteome database (2018 release). Approximately 1,000 proteins can be quantified with current methods.

Lipidomics analysis is performed according to state-of-the-art existing procedures and modified to apply the best available technology.

Chromatographic separation is performed on Waters Acquity BEH C18 column (1.7μm X 2.1mm X 100 mm) using the gradient of two standard mobile phases (mobile phase A contains water, 0.1% formic acid and 10 ml 1M ammonium acetate, mobile phase B composes isopropanol and acetonitrile (1:1) with the same addition of formic acid and ammonium acetate).

The Mass spectrometry identification of compounds is targeted based on a pre-made library of target metabolites in plasma.

Based on the results from the lipidomics analyses, we will select a panel of diagnostic markers, which will most efficiently describe the speed of the disease progression. For the selected biomarkers we will develop an absolute quantitative method, based on LC-MS-MS (triple quadrupole MS in MRM mode) methodology, using commercially available standard compounds, including stable isotope labelled compounds as internal standards.

The biological analysis and data management of proteomics and lipidomics will take place at the CBMR.

Transcriptomomics analyses To identify genes that play an important role in the progression or recompensation of AH, we will compare datasets from bulk RNA sequencing in AH to already established datasets from single cell RNS sequencing of the liver.

Based on genes that are simultaneously suggested by bulk-RNA in our samples and scRNAseq, we can explore the key transcriptional regulators in ALD.

We will make use of this resource to computationally deconvolute the bulk transcriptome data of the liver biopsies to estimate the relative abundance of each cell type of the liver (hepatocyte, hepatic stellate cells, liver sinusoidal epithelial cells, etc.) in each patient. Possible disease regulators of both progression and recompensation will be assessed.

All patients with a debut of AH, and irrespective of time and circumstances of diagnosis, comorbidities and severity of disease will be offered inclusion in the cohort. All participants will be engaged by either the physician or nurse providing standard of care. If they are interested in the study, all participants will be informed in writing as well as orally by study investigators and project nurses. All participants will be offered oral information about the study, and at least 24 hours of time for reflection before accepting inclusion. It will be emphasized that participation is voluntary and that the participant can withdraw at any time.

A proportion of patients will be diagnosed with severe AH where complications compromising their cognitive function, e.g. severe sepsis, hepatic encephalopathy or delirium is present. When complications are considered reversible, information and possible enrolment in the study will be delayed until the patient has recovered, but no more than two months from diagnosis. When complications are considered irreversible or there may be reasonable doubt of the patient's survival, patients will be considered eligible, but excluded to avoid unnecessary or unethical conduction of procedures.

The present study is an incidence-based cohort. When written consent based on oral and written information is obtained the patient will be enrolled in the trial.

For the study a research biobank will be established. The biobank will contain blood and stool collected at baseline, three months, and 12 months. If a participant has ascites and needs paracentesis, a subcutaneous fat biopsy will be taken from the incision spot on the abdomen.

The bio bank is registered by The Danish Data Protection Agency.

The direct benefits related to participation in the study is the motivation and support towards alcohol-cessation. There may be minor discomfort related to extra blood sampling. At twelve months, an extra procedure for transjugular liver-biopsy is conducted. Procurement of fat tissue biopsies are done in local anesthesia and only if participants are in need of paracentesis, which involves local anesthesia and perforation of skin and fat tissue on the abdomen.

The investigations of novel biomarkers and genomic variants are exploratory, and there is no direct benefit for the participants involved. There are no nuisance or disadvantage involved either. However, the project will provide novel information on risk associations in cirrhosis that may lead to new discoveries of therapeutic targets in AH. We therefore believe that the benefits of the study outweigh the disadvantages.

All results derived from the study will be sought published, irrespective of positive, negative or inconclusive nature. Listing of authors will follow the International Committee of Medical Journal Editors recommendations for authorship (ICMJE Vancouver guidelines).

The study will contribute to a better characterization of AH and contribute to an improved understanding of disease mechanisms in the future.

The study is initiated by medical physicians and nurses employed by the Gastro Unit, Universit Hospital Hvidovre.

The Novo Nordisk Foundation has supported the present study (NNF2024#0088416).

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of AH, supported by biochemistry (bilirubin 50 mmol/l or higher) and ultrasound or other imaging techniques.
* Informed written consent.

Exclusion Criteria:

* People where the diagnosis of AH is questioned with reasonable doubt.
* Withdrawal of informed consent.
* Persons eligible for inclusion where the investigational program is delayed or not initiated within two months after the diagnosis of suspected AH.
* Persons with hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the proteomic profile | 12 months
  Change from baseline to 12 months in the proteomic profile in the liver tissue
Change from baseline in the lipidomic profile | 12 months
  Changes from basline to 12 months in the lipidomic profile in the liver tissue
Number of participants in recompensation | 12 months
  Number of patients who achieve recompensation/remission from AH after 12 months

SECONDARY OUTCOMES:
Change in alcohol use from baseline | 12 months
  Change in alcohol use from baseline to 12 months by 30 days timeline followback.
Effect of motivational enhancement therapy | 3 months
  Number of participants who recieve motivational enhancement therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All data will be anonymized at the end of the trial and can be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2029-2034
Access Criteria: Proposals for data access will be evaluated in the study group.